CLINICAL TRIAL: NCT05270265
Title: A Phase Ia Study to Assess Safety and Immunogenicity of the Plasmodium Vivax Malaria Vaccine Candidate Pvs25-IMX313 in Matrix-M1 Adjuvant in Healthy Adults Living in the UK
Brief Title: Safety and Immunogenicity of Pvs25-IMX313/Matrix-M1 Vaccine
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to administrative delays in the approval of a substantial amendment to extend the shelf-life of Pvs25-IMX313. Regulatory approval was only received on 11 August 2023, after end of study visits had already been conducted.
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC084
Record Dates: First submitted 2022-01-28; First posted 2022-03-08 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2024-08

CONDITIONS: Malaria, Vivax
Keywords: Pvs25-IMX313; Matrix-M1
MeSH Terms: conditions — Malaria, Vivax | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (low dose) (Experimental): 8-10 volunteers receiving three doses of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pvs25-IMX313/Matrix-M1
- Group 2 (standard dose) (Experimental): 8-10 volunteers receiving three doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pvs25-IMX313/Matrix-M1
- Group 3 (fractional dose) (Experimental): 8-10 volunteers receiving two doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0 and 28, followed by one dose of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on day 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pvs25-IMX313/Matrix-M1

INTERVENTIONS:
Biological: Pvs25-IMX313/Matrix-M1 — Three doses of Pvs25-IMX313 in Matrix-M1 at different concentrations

SUMMARY:
This is an open-label, single-centre, non-randomised, first-in-human Phase Ia study to assess the safety and immunogenicity of the Pvs25-IMX313 vaccine, administered in Matrix-M1 adjuvant.

DETAILED DESCRIPTION:
Volunteers will be recruited into one of three groups (n=8-10 per group) at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford over approximately 18 months. All volunteers will receive three doses of Pvs25-IMX313 in Matrix-M1, administered intramuscularly and given four weeks apart. Enrolment will be staggered with clinical and safety reviews, follow-up visits and monitoring via a diary card.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their GP.
* Volunteers with the potential to become pregnant only: must practice continuous effective contraception for the duration of the study. Acceptable forms of contraception for volunteers of child-bearing potential are: Established use of oral, injected or implanted hormonal methods of contraception, Placement of an intrauterine device or intrauterine system, Male sterilization (if the vasectomised partner is the sole partner for the participant), True abstinence from sex with sperm-producing partners, when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence and withdrawal are not acceptable methods of contraception).
* Agreement to refrain from blood donation for the duration of the study.
* Able and willing to provide written informed consent to participate in the trial.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Use of immunoglobulins or blood products (e.g., blood transfusion) in the last three months.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination, with the exception of --COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination.
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Concurrent involvement in another clinical trial or planned involvement during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the -vaccine.
* Any history of anaphylaxis in reaction to vaccinations.
* Pregnancy, lactation or intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless volunteer has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV ribonucleic acid (RNA) PCR at screening for this study).
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in SOP VC027.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Vaccination and re-vaccination exclusion criteria:

Absolute contraindications:

* Anaphylactic reaction following administration of vaccine
* Pregnancy

Contraindications at that point in time (may be rescheduled):

* Acute disease (moderate/severe illness with or without fever)
* T>37.5C
* Current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR swab test taken during current illness or positive COVID-19 PCR swab or rapid antigen test within preceding 7 days without symptoms. Vaccinations will be delayed by a minimum of 7 days from the date of the first positive COVID-19 PCR swab or rapid antigen test, as long as symptoms are improving or resolved. It will be at the discretion of the Investigator to withdraw a participant if they develop severe COVID-19 disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, DPhil FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Low Dose): 8 volunteers receiving three doses of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
- Group 2 (Standard Dose): 9 volunteers receiving three doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
- Group 3 (Fractional Dose): 8 volunteers receiving two doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0 and 28, followed by one dose of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on day 56 via intramuscular injection (IM) in the deltoid region of the arm
Period: Overall Study
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Started | 8 | 9 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose) | Total
Number analyzed (Participants) | 8 | 9 | 8 | 25
Age, Customized [Median (Full Range); unit: years]
  Age | 29.5 [24 to 42] | 32 [23 to 40] | 27 [24 to 44] | 29 [23 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 3 | 4 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 4 | 5 | 4 | 13
  White Irish | 0 | 1 | 1 | 2
  White Other | 2 | 2 | 2 | 6
  Asian or Asian British | 1 | 0 | 0 | 1
  Black or Black British - African | 0 | 1 | 0 | 1
  Other Asian Background | 1 | 0 | 0 | 1
  Other - Latino | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Pvs25-IMX313/Matrix-M1 Vaccine in Healthy Adult Volunteers: Number of Participants Reporting Solicited Local Reactogenicity Signs and Symptoms
Description: Number of participants in each group who reported solicited local reactogenicity signs and symptoms in the 7 days following each vaccination. Solicited local reactogenicity signs and symptoms are collected through participant-reported e-diaries.
Time Frame: 7 days following each vaccination
Population: Percentages are the proportion of participants in each group that reported each symptom after at least one vaccination.
  Group 1: All participants received three vaccinations Group 2: 9 participants received vaccinations 1 and 2, 7 participants received vaccination 3 Group 3: 8 participants received vaccinations 1 and 2, 6 participants received vaccination 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Number analyzed (Participants) | 8 | 9 | 8
Participants
  Warmth: Mild | 1 | 3 | 3
  Warmth: Moderate | 0 | 0 | 0
  Warmth: Severe | 0 | 0 | 0
  Redness: Mild | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0
  Itch: Mild | 1 | 0 | 0
  Itch: Moderate | 0 | 0 | 0
  Itch: Severe | 0 | 0 | 0
  Pain: Mild | 8 | 7 | 5
  Pain: Moderate | 0 | 3 | 0
  Pain: Severe | 0 | 0 | 0

2. Primary Outcome: Safety and Tolerability of the Pvs25-IMX313/Matrix-M1 Vaccine in Healthy Adult Volunteers: Number of Participants Reporting Solicited Systemic Reactogenicity Signs and Symptoms.
Description: Number of participants in each group who reported solicited systemic reactogenicity signs and symptoms in the 7 days following each vaccination. Solicited systemic reactogenicity signs and symptoms are collected through participant-reported e-diaries.
Time Frame: 7 days following each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Number analyzed (Participants) | 8 | 9 | 8
Participants
  Arthralgia: Mild | 1 | 2 | 3
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Fatigue: Mild | 7 | 7 | 6
  Fatigue: Moderate | 1 | 4 | 2
  Fatigue: Severe | 0 | 0 | 1
  Myalgia: Mild | 2 | 4 | 5
  Myalgia: Moderate | 1 | 0 | 1
  Myalgia: Severe | 0 | 0 | 0
  Malaise: Mild | 3 | 4 | 5
  Malaise: Moderate | 1 | 0 | 3
  Malaise: Severe | 0 | 0 | 1
  Fever: Mild | 1 | 1 | 0
  Fever: Moderate | 1 | 0 | 1
  Fever: Severe | 0 | 0 | 0
  Feverishness: Mild | 2 | 4 | 4
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 1 | 1
  Nausea: Mild | 0 | 1 | 2
  Nausea: Moderate | 0 | 0 | 1
  Nausea: Severe | 0 | 0 | 0
  Headache: Mild | 6 | 3 | 5
  Headache: Moderate | 1 | 2 | 3
  Headache: Severe | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability of the Pvs25-IMX313/Matrix-M1 Vaccine in Healthy Adult Volunteers: Number of Unsolicited Adverse Events.
Description: Unsolicited adverse events were collected for 28 days following each vaccination through participant-reported e-diaries.
Time Frame: 28 days following each vaccination
Measure: Number; unit: Number of events
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Number analyzed (Participants) | 8 | 9 | 8
Number of events
  Total unsolicited adverse events (UAEs) | 56 | 54 | 53
  UAEs - no relationship to investigational vaccine | 26 | 20 | 14
  UAEs - unlikely related to investigational vaccine | 22 | 21 | 31
  UAEs - possibly related to investigational vaccine | 5 | 12 | 6
  UAEs - probably related to investigational vaccine | 3 | 1 | 2
  UAEs - definitely related to investigational vaccine | 0 | 0 | 0

4. Primary Outcome: Safety of the Pvs25-IMX313/Matrix-M1 Vaccine in Healthy Adult Volunteers: Occurrence of Abnormal Laboratory Test Results
Description: Occurrence of change from baseline laboratory test results
Time Frame: 28 days following vaccination
Measure: Number; unit: Number of abnormal laboratory results
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Number analyzed (Participants) | 8 | 9 | 8
Number of abnormal laboratory results
  Grade 1 laboratory abnormalities | 47 | 25 | 21
  Grade 2 laboratory abnormalities | 3 | 5 | 4
  Grade 3 laboratory abnormalities | 0 | 2 | 1

5. Primary Outcome: Safety and Tolerability of the Pvs25-IMx313/Matrix-M1 Vaccine in Healthy Adult Volunteers: Number of Serious Adverse Events
Description: Number of serious adverse events reported per group throughout the study period.
Time Frame: Whole duration of the study period (8 months following enrolment)
Measure: Number; unit: Number of serious adverse events
Arm/Group | Group 1 (Low Dose) | Group 2 (Standard Dose) | Group 3 (Fractional Dose)
Number analyzed (Participants) | 8 | 9 | 8
Number of serious adverse events | 0 | 0 | 0

6. Secondary Outcome: Humoral Immunogenicity of the Pvs25-IMX313/Matrix-M1 Vaccine When Administered to Healthy Adult Volunteers: Humoral Responses to the Pvs25 Protein
Description: Antibody responses to the Pvs25 protein will be assessed through total IgG isotypes and avidity
Time Frame: Days 1, 29, 57, 140 and 240.
Reporting Status: Not Posted

7. Secondary Outcome: Cellular Immunogenicity of the Pvs25-IMX313/Matrix-M1 Vaccine When Administered to Healthy Adult Volunteers: Cellular Responses to the Pvs25 Protein.
Description: T cell responses to Pvs25 will be assessed by ex vivo enzyme-linked immunospot assays (ELISpot) and flow cytometry assays.
Time Frame: Days 1, 29, 57, 140 and 240.
Reporting Status: Not Posted

8. Secondary Outcome: Ex Vivo Efficacy of the Pvs25-IMX313/Matrix-M1 Vaccine When Administered to Healthy Adult Volunteers: Transmission-Reducing Activity
Description: Transmission-reducing activity will be assessed through direct membrane feeding assays (DMFA).
Time Frame: Days 1, 29, 57, 140 and 240.
Reporting Status: Not Posted

9. Secondary Outcome: Ex Vivo Efficacy of the Pvs25-IMX313/Matrix-M1 Vaccine When Administered to Healthy Adult Volunteers: Transmission-Blocking Activity
Description: Transmission-blocking activity will be assessed through direct membrane feeding assays (DMFA).
Time Frame: Days 1, 29, 57, 140 and 240.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Solicited adverse event data was collected for 7 days post-vaccination. Unsolicited adverse event data was collected for 28 days post-vaccination.
Description: Solicited adverse events, along with severity and the number of participants affected per study group by each event, have been reported as part of the primary outcome measures.
Groups:
- Group 1: Low Dose: 8 volunteers receiving three doses of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
- Group 2: Mid Dose: 9 volunteers receiving three doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
- Group 3: Fractional Dose: 8 volunteers receiving two doses of 50 µg Pvs25-IMX313 in 50 µg Matrix-M1 on days 0 and 28, followed by one dose of 10 µg Pvs25-IMX313 in 50 µg Matrix-M1 on day 56 via intramuscular injection (IM) in the deltoid region of the arm
Arm/Group | Group 1: Low Dose | Group 2: Mid Dose | Group 3: Fractional Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Low Dose (N=8) | Group 2: Mid Dose (N=9) | Group 3: Fractional Dose (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Blocked nose (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (5)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Menstrual cramps/pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dog bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (4) | 1 (2)
Feverishness (Immune system disorders) | 0 (0) | 2 (3) | 0 (0)
Flu-like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gonorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (14) | 5 (8) | 4 (9)
Heartburn (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heatstroke (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Insect bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Iron-deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Irregular heartbeat (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Itch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
IUD complications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Joint ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Low mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 3 (4)
Migraine (General disorders) | 1 (8) | 0 (0) | 0 (0)
Mild eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Neck and shoulder ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pulled hamstring (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Immune system disorders) | 4 (4) | 1 (1) | 3 (3)
Rhinosinusitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sore neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 5 (10) | 5 (7)
Stomach ache/cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillar disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (General disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Whiplash (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Whooshing sound in one ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05270265/Prot_SAP_001.pdf